CLINICAL TRIAL: NCT06334380
Title: Virtual Reality for Surgical Prehabilitation and Rehabilitation
Brief Title: VR for Surgical Prehabilitation and Rehabilitation
Acronym: VR-PREP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cindy Kin, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 73688
Record Dates: First submitted 2024-03-14; First posted 2024-03-28 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Frailty; Surgery
Keywords: Prehabilitation; Rehabilitation; Virtual Reality; Physical Therapy; Breast Surgery; Breast Cancer; Breast Reconstruction; Axillary Surgery
MeSH Terms: conditions — Breast Neoplasms; Frailty

STUDY DESIGN:
Intervention Model Description: Participants randomized to one of two arms, VR self-paced modules with live PT guidance and VR without live PT guidance.
Who Masked: Outcomes Assessor
Masking Description: Blinded assessor will conduct adherence calls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Virtual Reality Modules Only (Active Comparator): Participants will have access to the prehabilitation (preoperative) and rehabilitation (postoperative) virtual reality physical therapy modules.
  Interventions: Other: Virtual Reality Modules Only
- Intervention Group: Virtual Reality Modules + Live Physical Therapist Support (Experimental): Participants will have access to prehabilitation and rehabilitation virtual reality physical therapy modules in addition to zoom "office hours" with the physical therapist so that they may ask questions.
  Interventions: Other: Virtual Reality Modules + Live Physical Therapist Support

INTERVENTIONS:
Other: Virtual Reality Modules Only — Participants will complete self-paced VR modules prior to and after surgery (prehab/rehab) and will be provided with technical assistance from the study team.
  Arms: Control Group: Virtual Reality Modules Only
Other: Virtual Reality Modules + Live Physical Therapist Support — Participants will complete self-paced VR modules prior to and after surgery (prehab/rehab) and will be provided with technical assistance from the study team. Participants will also have access to up to three live PT sessions via Zoom where they can ask questions and complete modules with PT feedback.
  Arms: Intervention Group: Virtual Reality Modules + Live Physical Therapist Support

SUMMARY:
This randomized controlled trial aims to determine feasibility and acceptability of of VR-physical therapy modules for surgical patients undergoing breast or axilla surgery in order to prepare for and recover from surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* English speaking
* Will undergo breast or axilla surgery at Stanford
* Have access to internet and stable Wifi at home
* Have access to a space with stable chair at home
* Ability to sit-to-stand without significant balance issues
* Absence of chronic vertigo or nausea/vomiting
* Agreeable to up to 4 weeks of prehab prior to surgery and up to 8 weeks of post-operative rehab

Exclusion Criteria:

* Inability to engage in PT due to physical limitations identified by the participant and/or care team
* Inability to complete a brief online survey at three time points during the duration of the study
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
VR for remote Physical Therapy (PT) | 12 weeks
  This study will evaluate the feasibility of using VR technology to perform PT remotely from patients' homes to prepare for and recover from surgery. Frequency of engagement with the VR system (e.g., number of times participant initiated a VR physical therapy module, how long each session was used for) will be measured. Engagement with the live PT sessions will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No